CLINICAL TRIAL: NCT01977521
Title: Transcranial Direct Current Stimulation as Treatment for Auditory Hallucinations A Sham-controlled Trial
Brief Title: Transcranial Direct Current Stimulation as Treatment for Auditory Hallucinations
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iris Sommer (Other)
Responsible Party: Sponsor-Investigator, Iris Sommer, Professor, Psychiatrist, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS_UMC
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Psychotic Disorders; Mood Disorders; Personality Disorders; Stress Disorders, Post-Traumatic; Hearing Disorders
MeSH Terms: conditions — Psychotic Disorders; Mood Disorders; Personality Disorders; Stress Disorders, Post-Traumatic; Hearing Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): transcranial direct current stimulation (2mA)
  Interventions: Device: Eldith DC Stimulator stimulation
- Sham (Sham Comparator): Sham stimulation
  Interventions: Device: Eldith DC Stimulator sham stimulation

INTERVENTIONS:
Device: Eldith DC Stimulator stimulation — The anodal electrode will be placed with the middle of the electrode over a point midway between F3 and FP1 (left prefrontal cortex: dorsolateral prefrontal cortex and the cathodal electrode located over a point midway between T3 and P3 (left temporo-parietal junction). Stimulation will consist of 2 mA for 20 minutes per session.
  Arms: Treatment
Device: Eldith DC Stimulator sham stimulation — The anodal electrode will be placed with the middle of the electrode over a point midway between F3 and FP1 (left prefrontal cortex: dorsolateral prefrontal cortex and the cathodal electrode located over a point midway between T3 and P3 (left temporo-parietal junction). In the sham condition, after 40 seconds of real stimulation (2 mA), only a small current pulse will occur every 550 msec (110 mA over 15 msec) through the remainder of the 20-minute period.
  Arms: Sham

SUMMARY:
The present study aims to examine the efficacy of transcranial direct current stimulation on the severity of auditory hallucinations.

DETAILED DESCRIPTION:
Rationale: Auditory hallucinations (AH) are a symptom of several psychiatric disorders, such as schizophrenia. In the majority of patients, these AH respond well to antipsychotic medication. Yet, a significant minority continues to experience frequent AH despite optimal pharmacotherapy and AH severely decrease quality of life in these patients. The number of alternative treatment options for this medication resistant group is currently low and most of them focus on coping with the hallucinations. Transcranial direct current stimulation (tDCS), in contrast, is a safe, non-invasive technique that is able to directly influence cortical excitability through the application of very low electric currents. This technique has only a few transient side-effects and is cheap and portable. To date, only one randomized controlled trial has been published, suggesting high efficacy of tDCS for the treatment of medication-resistant AH in a relatively small sample. We aim to replicate and extend these findings by investigating the efficacy of this technique in a larger sample.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18.
* Frequent auditory hallucinations (at least 5 times a week).
* Patients are on a stable dose of antipsychotic medication (which can also be zero) for at least 2 weeks
* Mentally competent for informed consent.
* Provided informed consent.

Exclusion Criteria:

* Metal objects in or around the head that cannot be removed (i.e. cochlear implant, surgical clips, piercing)
* History of seizures, or a history of seizures in first-degree relatives.
* History of eye trauma with a metal object or professional metal workers
* History of brain surgery, brain infarction, head trauma, cerebrovascular accident, broken skull, brain tumour, heart disease, cardiac pacemaker.
* Skin disease on the scalp on the position of the tDCS electrodes
* Coercive treatment based on a judicial ruling
* Pregnancy in female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Total score of the Auditory Hallucination Rating Scale (AHRS) questionnaire | 4 years
  The primary outcome is the change in the severity of the hallucinations before and after the treatment, as experienced by the participant, measured with the Auditory Hallucination Rating Scale (AHRS)

SECONDARY OUTCOMES:
Changes in severity of hallucinations as assessed by the hallucination change scale (HCS)questionnaire | 4 years
Changes of positive, negative and disorganized symptomatology as assessed by the positive and negative syndrome scale (PANSS) | 4 years
Severity of psychotic symptoms will be measured by the questionnaire for psychotic symptoms (QPS) | 4 years
Prior expectations regarding the efficacy of the treatment of the participants | 4 years
Strength of the motor threshold as assessed using TMS | 4 years
The presence and severity of side-effects will be monitored using the tDCS adverse effects questionnaire | 4 years
Interference score on the Stroop task | 4 years
Score on the Trailmaking test A and B | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Iris Sommer, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC, Utrecht, Netherlands

REFERENCES:
- [Derived] Koops S, Blom JD, Bouachmir O, Slot MI, Neggers B, Sommer IE. Treating auditory hallucinations with transcranial direct current stimulation in a double-blind, randomized trial. Schizophr Res. 2018 Nov;201:329-336. doi: 10.1016/j.schres.2018.06.010. Epub 2018 Jun 20. PMID 29934249